CLINICAL TRIAL: NCT05950282
Title: Measuring Fasting Insulin and HOMA-IR by Age, Sex, Race/Ethnicity, BMI, and PCOS Diagnosis
Brief Title: Fasting Insulin and HOMA-IR by Age, Sex, Race/Ethnicity, BMI, and PCOS Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Lilli Health (Other)
Responsible Party: Principal Investigator, Ali Chappell, Founder and CEO, Lilli Health
Other Study IDs: 2023-0060
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Insulin Resistance; Polycystic Ovary Syndrome; Hyperinsulinism; Obesity; Metabolic Syndrome
Keywords: PCOS; Hyperinsulinemia; Insulin Resistance; Metabolic Syndrome; Obesity; Type 2 Diabetes
MeSH Terms: conditions — Insulin Resistance; Polycystic Ovary Syndrome; Hyperinsulinism; Obesity; Metabolic Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study aims to investigate the relationship between fasting insulin and Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) across various demographic factors, including age, sex, race/ethnicity, BMI, and polycystic ovary syndrome (PCOS) diagnosis. By analyzing these variables, the study seeks to identify potential variations in insulin levels, which could provide valuable insights into the impact of different factors on metabolic health and the development of insulin-related conditions.

DETAILED DESCRIPTION:
This study aims to investigate the significance of measuring fasting insulin and the homeostatic model assessment of insulin resistance (HOMA-IR) in identifying metabolic health across various demographic and clinical factors. Specifically, the study will examine the influence of age, sex, race/ethnicity, BMI, and polycystic ovary syndrome (PCOS) diagnosis on insulin levels and insulin resistance as essential indicators of metabolic dysfunction.

Metabolic health disorders, such as insulin resistance and impaired glucose metabolism, are known to be associated with an increased risk of developing conditions like type 2 diabetes, cardiovascular diseases, and metabolic syndrome. Traditionally, glucose levels have been used to assess metabolic health; however, fasting insulin and HOMA-IR provide valuable insights into the underlying insulin dysregulation that precedes the onset of these conditions.

Disparities in insulin levels have been observed across different racial and ethnic groups. These variations may arise from genetic predispositions, differences in lifestyle, or a combination of both, thus highlighting the need to explore these factors comprehensively. BMI, a measure of body composition, has been strongly associated with elevated insulin levels and insulin resistance. Individuals with obesity often exhibit dysregulated insulin metabolism, leading to higher fasting insulin and HOMA-IR values. Furthermore, PCOS, a common endocrine disorder affecting reproductive-age women, is frequently associated with insulin resistance. Studying the insulin profiles among women with PCOS will shed light on the potential metabolic implications and help tailor interventions for this at-risk population.

The study will employ a cross-sectional design, enrolling a large sample of participants from diverse backgrounds. Fasting insulin levels will be measured using standardized laboratory methods, and HOMA-IR scores will be calculated based on fasting insulin and glucose values. Statistical analyses, including regression models and subgroup comparisons, will be conducted to assess the associations between fasting insulin, HOMA-IR, and the demographic and clinical factors of interest.

This research aims to emphasize the importance of incorporating fasting insulin and HOMA-IR measurements alongside glucose assessments to enhance the identification and understanding of metabolic health disorders. The findings are expected to contribute to a more comprehensive approach in diagnosing, managing, and preventing metabolic diseases, ultimately leading to improved patient outcomes and public health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants aged 18+ years.
* Sex: Both males and females.
* Race/Ethnicity: Participants from diverse racial and ethnic backgrounds
* BMI: Participants with a range of body mass index (BMI) values
* PCOS Diagnosis: Participants with and without a confirmed diagnosis PCOS based on established diagnostic criteria.

Exclusion Criteria:

* Age: Participants below 18 years
* Sex: None. Both males and females are included.
* Race/Ethnicity: None. Participants from all racial and ethnic backgrounds are included.
* Endocrine Disorders: Participants with other endocrine disorders affecting insulin levels, such an insulin secreting tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to investigate the levels of Fasting Insulin and HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) among individuals with varying characteristics, including age, sex, race/ethnicity, BMI (Body Mass Index), and PCOS (Polycystic Ovary Syndrome) diagnosis. The study population consists of a diverse group of participants referred by healthcare providers and online platforms to purchase at-home insulin and HOMA-IR testing kits from the lillihealth.com website.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Fasting Insulin levels and HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) scores among different groups stratified by age, sex, race/ethnicity, BMI, and PCOS (Polycystic Ovary Syndrome) diagnosis. | 3 years
  The primary objective is to investigate the association between these measures and the specified demographic and clinical factors, providing insights into the variations and potential disparities in insulin resistance across different subgroups.

SECONDARY OUTCOMES:
Identify any significant interactions or relationships between the primary outcomes (Fasting Insulin and HOMA-IR) and the demographic and clinical factors, including age, sex, race/ethnicity, BMI, and PCOS diagnosis. | 3 years
  The secondary outcome measure will provide a comprehensive understanding of how various factors may influence insulin resistance and contribute to its heterogeneity in different populations.

CONTACTS AND LOCATIONS:
Overall Officials: Ali M Chappell, Principal Investigator — Lilli Health
Locations (1):
- Lilli Health, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lilli Health Website — https://www.lillihealth.com